CLINICAL TRIAL: NCT04439422
Title: Short Structured Psychological Intervention for Adults With ADHD - a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cereb AB (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Berkeh Nasri, PhD, Head of Research and Development, Cereb AB
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAINT
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Attention Deficit; Psychological Intervention; CBT; DBT; Self-Help; Adherence; Short Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAINT (Experimental)
  Interventions: Behavioral: Short ADHD Intervention
- Self-help material (Active Comparator)
  Interventions: Other: Self-help material with limited therapist support

INTERVENTIONS:
Behavioral: Short ADHD Intervention — Short, intensive psychological intervention based on CBT and DBT practices
  Other Names: SAINT
  Arms: SAINT
Other: Self-help material with limited therapist support — Self-help material from an evidence-based treatment manual for adult ADHD with access to limited therapist support via Internet (control group)
  Arms: Self-help material

SUMMARY:
The purpose of this study is to evaluate the effects of a novel psychological intervention for adult ADHD through a randomized controlled trial. Participants will be randomized to receive either a face-to-face manualized short psychological intervention, SAINT, or corresponding self-help material with limited access to therapist support. The main objective is to evaluate whether SAINT will show better outcomes on measures of ADHD-related symptoms, everyday function, and quality-of-life measures, when compared to the self-help material, and if any possible differences in outcomes are related to better treatment adherence in SAINT.

DETAILED DESCRIPTION:
ADHD is associated with deficiencies in short-term memory and executive function, negatively affecting patients' abilities to organize, schedule, multitask, follow through on instructions and finish jobs. This leads to uneven performance and possibly chronic underperformance in relation to actual intellectual resources. Psychiatric comorbidity is common for patients with ADHD, with 70-80% of adult patients meeting the criteria for at least one more clinical diagnosis. ADHD is also associated with sensation seeking and reckless behavior, including substance use and criminal activity.

Despite an increase in demand for assessment and treatment of ADHD among adults, access to evidence-based treatment is limited. In Sweden, most adult patients with ADHD are only offered pharmacological treatment. Pharmacological treatment, while in many cases effective, does not meet the demands of all patients, with 20-50% of patients not experiencing enough initial effect and/or excessive side-effects. Pharmacological treatment of ADHD also shows problems with long-term adherence, with approximately half of patients terminating treatment within the first two years, regardless of initial effect. Research on psychological treatment for adult ADHD is limited, though studies on behavioral treatment, including short-term therapies based on cognitive behavior therapy (CBT) and dialectic behavior therapy (DBT), have shown promising results.

This project, dubbed Short ADHD Intervention (SAINT), is based on previous research and pilot-studies of psychological treatments for adult ADHD. An existing treatment manual, based on CBT and DBT practices, will be fitted into a five-session, intensive face-to-face behavioral intervention, with a booster session at a one-month follow-up. The intervention will be compared to an equally long, active comparative control, consisting of self-help material and limited therapist support via Internet. Approximately 80 participants will be recruited at outpatient clinics in Stockholm. The participants will be randomized to receive either SAINT or the self-help material and limited therapist support.

ELIGIBILITY:
Inclusion Criteria:

* Swedish citizen
* Clinical Diagnosis of ADHD according to DSM-IV or DSM-5.
* Score of 17 or higher on the Adult ADHD Self Report Scale (ASRS v1.1), on any one of the two subscales.
* Not medically treated for ADHD symptoms throughout the study period, or medically treated with central stimulants or comparable substances since at least one month, with no significant changes in dosage and no anticipated significant changes in dosage.
* No change in any other medical treatment for psychiatric symptoms.
* Ability to participate in treatment during the study period.
* Abstinence from illegal substance use for at least three months.
* Access to and ability to use Internet and mobile phone during the study period.
* Ability to understand Swedish in speech and writing, and ability to fill-out forms online.

Exclusion Criteria:

* Clinical diagnosis of substance use disorder within three months prior to screening. Earlier episodic use of illegal substances is not excluding.
* Co-existing psychiatric condition or disorder expected to render the participant unable to follow-through the study processes.
* IQ ≤85 according to a prior neuropsychological assessment.
* Suicidality assessed at the first assessment interview.
* Organic brain syndrome.
* Autism spectrum disorder (ASD) where function is deemed too low for the treatment to be carried out, defined as ASD level 2 and level 3 according to DSM-5 and/or ASD with accompanying intellectual impairment and/or accompanying language impairment.
* Severe depression, defined as >34 on the MADRS-S or at a clinical assessment.
* Other current psychological treatment for ADHD or prior participation in treatment deemed to interfere with the study design.
* Limited or very limited self-rated recognition of problems regarding impulse control and/or emotional instability, in combination with low self-rated impairment, on a tailor-made measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change (from baseline) on The Adult ADHD Quality of Life Questionnaire (AAQoL) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)

SECONDARY OUTCOMES:
Change (from baseline) on ADHD Self-Report Scale (ASRS; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on the ADHD Rating Scale (ADHD RS; Assessed by an expert rater) | Baseline, 5 weeks (post treatment)
Change (from baseline) on Montgomery Åsberg Depression Rating Scale (MADRS-S; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on Sheehan Disability Scale (SDS; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on Difficulties in Emotion Regulation Scale (Brief Version; DERS-16; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on Satisfaction With Life Scale (SWLS; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on Perceived Stress Scale (PSS; Self-report) | Baseline, 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
Change (from baseline) on Clinical Global Impression - Severity Scale (CGI-S; Assessed by an expert rater) | Baseline, 5 weeks (post treatment)

OTHER OUTCOMES:
Clinical Global Impression - Improvement Scale (CGI-I; Assessed by an expert rater) | 5 weeks (post treatment)
Client Satisfaction Questionnaire (CSQ-8; Self-report) | 5 weeks (post treatment)
Treatment Credibility Scale (TCS; Self-report) | 1 week, 3 weeks
Treatment Evaluation (Self-report) | 5 weeks (post treatment)
  A tailor-made formulary to evaluate the participants' experience of the interventions, including any possible difficulties.
Adherence to Treatment (Self-report) | 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks (post treatment),9 weeks (FU1) 17 weeks (FU3)
  Using a tailor-made formulary.
Session Attendance (Assessed by an expert rater) | 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks (post treatment), 9 weeks (FU1)
  SAINT arm only.
Adverse Events During Treatment (Self-report) | 5 weeks (post treatment), 9 weeks (FU1) 17 weeks (FU3)
  Using a tailor-made formulary.
Changes in Other Treatment(s) During the Study Period (Self-report) | 5 weeks (post treatment),9 weeks (FU1) 17 weeks (FU3)
  Using a tailor-made formulary.

CONTACTS AND LOCATIONS:
Locations (1):
- Cereb AB, Stockholm, Sweden